CLINICAL TRIAL: NCT00159887
Title: A Multi-Centre, Multinational, Long-Term Extension Study, to Assess the Safety and Toleration of Subject Optimised Treatment Regimens of Oral Sildenafil Citrate for Pulmonary Arterial Hypertension in Subjects Who Have Completed Study A1481140.
Brief Title: Study to Assess the Longterm Safety of Sildenafil Citrate in Patients With Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1481142
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil citrate

SUMMARY:
Open label extension study to the pivotal efficacy study to assess the safety of sildenafil citrate in patients with pulmonary arterial hypertension

ELIGIBILITY:
Inclusion Criteria:

* Patients with PAH who had completed the 12 week pivotal study

Exclusion Criteria:

* Any other patients with PAH that had not been included into the pivotal study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2002-12; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Safety
Standard safety data
Efficacy
6-Minute Walk Test
BORG Dyspnoea Score
WHO Functional Class
Quality of Life SF-36 and EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (54):
- United States (16):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Australia (2):
  - Pfizer Investigational Site, Darlinghurst, New South Wales
  - Pfizer Investigational Site, Melbourne, Victoria
- Belgium (2):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Leuven
- Pfizer Investigational Site, São Paulo, São Paulo, Brazil
- Pfizer Investigational Site, Prague, Czechia
- Pfizer Investigational Site, Copenhagen, Denmark
- Pfizer Investigational Site, Clamart, France
- Germany (3):
  - Pfizer Investigational Site, Giessen
  - Pfizer Investigational Site, Hanover
  - Pfizer Investigational Site, Leipzig
- Pfizer Investigational Site, Shatin NT, Hong Kong
- Hungary (2):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Zalaegerszeg
- Israel (2):
  - Pfizer Investigational Site, Petah Tikva
  - Pfizer Investigational Site, Tel Litwinsky
- Italy (2):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Pisa
- Malaysia (2):
  - Pfizer Investigational Site, Kuala Lumpur
  - Pfizer Investigational Site, Petaling Jaya
- Mexico (2):
  - Pfizer Investigational Site, Tlalpan Mexico, Mexico City
  - Pfizer Investigational Site, Tlalpan, Mexico DF
- Pfizer Investigational Site, Amsterdam, Netherlands
- Poland (2):
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Zabrze
- Pfizer Investigational Site, Singapore, Singapore
- South Africa (3):
  - Pfizer Investigational Site, Parow, Western Cape
  - Pfizer Investigational Site, Parktown
  - Pfizer Investigational Site, Parktown West
- Pfizer Investigational Site, Suwon, South Korea
- Spain (2):
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
- Pfizer Investigational Site, Gothenburg, Sweden
- United Kingdom (5):
  - Pfizer Investigational Site, Papworth Everard, Cambridgeshire
  - Pfizer Investigational Site, Sheffield, South Yorkshire
  - Pfizer Investigational Site, Newcastle upon Tyne, Tyne and Wear
  - Pfizer Investigational Site, Cambridge
  - Pfizer Investigational Site, Glasgow

REFERENCES:
- [Derived] Wirostko BM, Tressler C, Hwang LJ, Burgess G, Laties AM. Ocular safety of sildenafil citrate when administered chronically for pulmonary arterial hypertension: results from phase III, randomised, double masked, placebo controlled trial and open label extension. BMJ. 2012 Feb 21;344:e554. doi: 10.1136/bmj.e554. PMID 22354598
- [Derived] Rubin LJ, Badesch DB, Fleming TR, Galie N, Simonneau G, Ghofrani HA, Oakes M, Layton G, Serdarevic-Pehar M, McLaughlin VV, Barst RJ; SUPER-2 Study Group. Long-term treatment with sildenafil citrate in pulmonary arterial hypertension: the SUPER-2 study. Chest. 2011 Nov;140(5):1274-1283. doi: 10.1378/chest.10-0969. Epub 2011 May 5. PMID 21546436
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481142&StudyName=Study%20to%20Assess%20%20the%20Longterm%20Safety%20of%20Sildenafil%20Citrate%20in%20Patients%20with%20Pulmonary%20Arterial%20Hypertension